CLINICAL TRIAL: NCT00857168
Title: A Phase I Trial to Determine the Impact of Application of Antiperspirant and Deodorant as Well as Washing the Application Site, on the Pharmacokinetics of Testosterone Following Single Dose Applications of 2% Testosterone MD-Lotion® (Cutaneous Solution)
Brief Title: To Determine the Effects of Deodorant, Antiperspirant and Washing on the Pharmacokinetics of 2% Testosterone MD Lotion
Acronym: MTE10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrux DDS Pty Ltd (Industry)
Responsible Party: Tina Soulis, Director, CLinical Devleopment, Acrux Pharma Pty Ltd
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MTE10
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Active Comparator)
  Interventions: Drug: Testosterone MD-Lotion
- Group 2 (Active Comparator)
  Interventions: Drug: Testosterone MD-Lotion
- Group 3 (Active Comparator)
  Interventions: Drug: Testosterone MD-Lotion
- Group 4 (Active Comparator)
  Interventions: Drug: Testosterone MD-Lotion
- Group 5 (Active Comparator)
  Interventions: Drug: Testosterone MD-Lotion
- Group 6 (Active Comparator)
  Interventions: Drug: Testosterone MD-Lotion

INTERVENTIONS:
Drug: Testosterone MD-Lotion

SUMMARY:
Testosterone replacement treatment is the most effective way of treating hypogonadism in men.

Acrux has a propriety testosterone replacement product, Testosterone MD-Lotion and this study will evaluate the impact of application of antiperspirant and deodorant on absorption of testosterone, when applied pre-application of Testosterone MD-Lotion® (cutaneous solution).

The study also aim to evaluate the impact of washing the application site on the absorption of testosterone, when washed post-application of Testosterone MD-Lotion® (cutaneous solution).

ELIGIBILITY:
Inclusion Criteria:

* Healthy premenopausal female subjects ≥18 and ≤45 years of age with qualifying general medical health.

Exclusion Criteria:

* Disqualifying concurrent condition or allergy/sensitivity to testosterone replacement therapy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of application of antiperspirant and deodorant on absorption of testosterone, when applied pre-application of Testosterone MD-Lotion® (cutaneous solution). Also to evaluate the impact of washing. | April 2009

SECONDARY OUTCOMES:
To assess the safety and tolerability of Testosterone MD-Lotion® (cutaneous solution) following single dose application. | April 2009

CONTACTS AND LOCATIONS:
Overall Officials: Tina Soulis, PhD, Study Director — Acrux Pharma Pty Ltd
Locations (1):
- QPharm Pty Ltd, Brisbane, Queensland, Australia